CLINICAL TRIAL: NCT07384312
Title: Study on the Antidepressant Effects and Mechanism of Action of Cang-ai Volatile Oil Based on Near-Infrared Functional Brain Imaging and the NT-Trk Signalling Pathway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dongdong Qin (Other)
Responsible Party: Sponsor-Investigator, Dongdong Qin, Researcher, Yunnan University of Chinese Medicine
Organization: Yunnan University of Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: XS2022-015
Record Dates: First submitted 2026-01-19; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Depression Disorder

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind controlled trial was conducted with 60 eligible patients, evenly divided by gender into an experimental group and a control group, with 30 patients in each. The experimental group received inhalation therapy with CAVO, while the control group received inhalation of bergamot essential oil. Both groups inhaled one drop (0.05 ml per drop) of 10% concentration of either Artemisia capillaris volatile oil or bergamot essential oil via a dropper inserted into a perfume diffuser, which was secured near the nasal area of the mask with a magnet. Participants were instructed to continuously sniff for 1 hour daily. Blood pressure, heart rate, anxiety, depression, and sleep scale scores were measured before and after inhalation. Serum levels of cortisol, IL-1, IL-2, IL-6, and TNF-α were quantified to assess biochemical changes. Functional near-infrared spectroscopy (fNIRS) was used to measure the relative concentrations of oxyhemoglobin and deoxyhemoglobin in the cerebral
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAVO group (Active Comparator): The experimental group received CAVO inhalation therapy, with 0.05 ml (1 drop) of 10% Artemisia absinthium volatile oil dripped into the aroma diffusion capsule using a Pasteur pipette. The capsule was secured near the participant's nose on the mask with a magnet, and they were instructed to continue inhaling continuously for 1 hour daily.
  Interventions: Drug: Cang-ai Volatile Oil
- BEO Group (Active Comparator): The control group received BEO inhalation therapy, with one drop (0.05 ml) of 10% bergamot essential oil instilled into the aroma diffuser bottle using a Pasteur pipette. The diffuser was secured near the nasal area of the mask with a magnet, and participants were instructed to continuously sniff the aroma for one hour daily.
  Interventions: Drug: Bergamot Essential Oil

INTERVENTIONS:
Drug: Cang-ai Volatile Oil — The experimental group received CAVO inhalation therapy, during which one drop (0.05 ml) of 10% mugwort volatile oil was administered into the aromatherapy diffuser using a Pasteur pipette. The diffuser was secured near the participant's nose on the mask with a magnet, and subjects were instructed to continuously inhale for one hour each day.
  Arms: CAVO group
Drug: Bergamot Essential Oil — The control group received BEO inhalation therapy, during which one drop (0.05 mL per drop) of 10% mandarin essential oil was administered into the aroma diffuser using a Pasteur pipette. The diffuser was secured near the participant's nose with a magnet fixed to the mask. Participants were instructed to continue smelling the aroma for 1 hour daily.
  Arms: BEO Group

SUMMARY:
This project plans to recruit 60 patients with depression, randomly assigning them to either the CAVO group or the bergamot essential oil group, with 30 participants in each. Quantitative measurement will be conducted using fNIRS technology to assess the impact of the intranasal CAVO pathway on brain functional connectivity during rest and brain activation during task performance. The antidepressant effects of CAVO will be evaluated using standardized depression scales, and target brain regions for CAVO's action will be identified through this process.

ELIGIBILITY:
Inclusion：

1. Meets the diagnostic criteria for depressive episodes as outlined in the fifth edition (revised) of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
2. Meets the diagnostic criteria for depression syndrome as defined in Part 1: Diseases of the Terminology for Clinical Diagnosis and Treatment in Traditional Chinese Medicine, issued by the National Administration of Traditional Chinese Medicine in 2023.
3. Scores on the 21-item Beck Depression Inventory (BDI) range from 10 to 15; scores on the 24-item Hamilton Depression Rating Scale (HAMD) range from 8 to 20.
4. Has a normal olfactory function, no history of allergic or respiratory diseases, aged 18-26 years.
5. At least one week prior to assessment, has not used antidepressants, other psychotropic medications, electroconvulsive therapy, or undergone transcranial magnetic stimulation or other physical therapies.
6. Exhibits depressive symptoms persisting for more than two weeks.
7. Right-handed.
8. Approved by the hospital ethics committee; all participants volunteer and have provided written informed consent.

Exclusion ：

1. Strict exclusion of individuals with a history of schizophrenia, alcohol dependence, or substance abuse.
2. Presence of organic brain disease, endocrine disorders, or depression secondary to other mental illnesses.
3. A score of ≥3 points on the suicidal item of the Hamilton Depression Rating Scale.
4. Pregnant or lactating women, or those with a history of manic or hypomanic episodes.
5. Family history of monomorphic or bipolar affective disorder.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Monitoring the relative concentration changes of oxyhemoglobin (HbO₂) and deoxyhemoglobin (deoxy-Hb) in cortical regions such as the frontal lobe, temporal lobe, and parietal lobe during near-infrared spectroscopy (NIRS) brain functional imaging. | From enrollment to the completion of one month of treatment
  Prior to the experiment, near-infrared brain functional imaging was conducted during resting and task states. Participants were provided with aromatherapy clips infused with either Mugwort volatile oil or Bergamot essential oil and instructed to smell the oils daily for one hour. After one month of this routine, follow-up near-infrared functional imaging was performed during resting and task conditions.

SECONDARY OUTCOMES:
Complete the questionnaire. | From enrollment to the completion of one month of treatment
  A baseline assessment was conducted using the Beck Depression Inventory prior to the commencement of the experiment, with a follow-up assessment performed one month later using the same standardised scale to evaluate changes in the severity of depression. The BDI-II scale ranges from 0 to 63 points, with diagnostic significance assigned to each score range as follows: 0-13 points: No depression or very mild depression 14-19 points: Mild depression 20-28 points: Moderate depression 29-63 points: Severe depression
Complete the questionnaire. | From enrollment to the completion of one month of treatment
  A baseline assessment was conducted using the Hamilton Depression Scale prior to the commencement of the experiment, with a follow-up assessment performed one month later using the same standardised scale to evaluate changes in the severity of depression. The HAMD-24 scale ranges from 0 to 96 points, with diagnostic significance assigned to each score band as follows: 0-7 points: Normal; 8-20 points: Possible depression; 21-34 points: Confirmed depression; 35-96 points: Severe depression

CONTACTS AND LOCATIONS:
Locations (1):
- Yunnan University of Chinese Medicine, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No
No consent for IPD sharing was obtained from participants.